CLINICAL TRIAL: NCT01043315
Title: Cognitive Function in Adults With Cardiac Disease
Acronym: TimePoints
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Richard Josephson, MS MD, Professor of Medicine, University Hospitals Cleveland Medical Center
Other Study IDs: 05-09-25
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Cognitive Impairment; Cardiac Disease
Keywords: Cognitive Function; Cognitive Impairment; Hospitalization; Cardiac Disease
MeSH Terms: conditions — Cognitive Dysfunction; Heart Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hospitalized Cardiac Patient: Adults admitted to Coronary intensive unit being treated for acute cardiovascular conditions

SUMMARY:
The purpose of this study is to identify cardiac patients' degree of unappreciated mild impairment in cognitive function patterns of cognitive function, and influencing factors related to cognitive functioning during hospitalization. The results from the study will contribute to tailoring the delivery of patient education to optimize patient understanding of information in future clinical practice.

It is hypothesized that the study will demonstrate the following:

1. The degree of cognitive function for patients hospitalized in a CICU will be below the scores for normal functioning adults.
2. Patients with acute cardiovascular conditions will score differently in cognitive functioning at various times throughout their hospitalization.
3. Relationships between cognitive function and following variables:

   * Patients with greater sleep deprivation or fatigue will exhibit lower cognitive functioning.
   * Patients with greater hunger will exhibit lower cognitive functioning.
   * Patients who are experiencing greater anxiety will exhibit lower cognitive functioning.
   * Patients who are experiencing depression will exhibit lower cognitive functioning.
   * Patients who have undergone or will undergo shortly treatment or procedures will exhibit lower cognitive functioning.

ELIGIBILITY:
Inclusion Criteria:

* Admission to the Cardiac Intensive Care Unite for acute cardiological issues during time of enrollment.
* Patients with NYHA class I, II, III, and IV.
* 18 years or older and must be awake and conversant at time of enrollment.

Exclusion Criteria:

* History of neurological disorder or injury (e.g., Alzheimer's Disease, dementia, stroke, seizures).
* Moderate or severe head injury (defined as > 24 hours loss of consciousness)
* Past or current history of severe psychiatric illness. Specifically, psychotic disorders (e.g., schizophrenia) and bipolar disorder. Potential participants will not be excluded on the basis of managed depression or anxiety disorder. These conditions are common in cardiac patients and their exclusion may limit the generalizability of findings.
* 5 years past or current history of alcohol or drug abuse (defined by DSM-IV criteria).
* History of learning disorder or developmental disability (defined by DSM-IV criteria).
* Renal failure requiring dialysis.
* History of sleep apnea (defined through previous sleep studies).
* Severely ill individuals, including those who are sedated, on a ventilator, exhibiting acute hemodynamic changes, and/or those deemed inappropriate by patient's physician to participate in study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients hospitalized in the University Hospitals' (Cleveland, OH) coronary intensive unit (CICU) being treated for acute cardiovascular conditions
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Cognitive Function as measured by Modified Mini Mental Status (3MS) Examination | Up to 3 hours prior to discharge
Cognitive Function as measured by Rey Auditory Verbal Learning | Up to 3 hours prior to discharge
Cognitive Function as measured by Trails testing | Up to 3 hours prior to discharge
Cognitive Function as measured by Digit Span Backwards | Up to 3 hours prior to discharge
Cognitive Function as measured by Rey Auditory Verbal Learning Long Delay | Up to 3 hours prior to discharge
Cognitive Function as measured by Rey Auditory Verbal Learning Long Delay and Recognition | Up to 3 hours prior to discharge
Cognitive Function as measured by Frontal Assessment Battery | Up to 3 hours prior to discharge

CONTACTS AND LOCATIONS:
Overall Officials: Richard Josephson, MS, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals of Cleveland, Cleveland, Ohio, United States